CLINICAL TRIAL: NCT00652769
Title: A Randomized Controlled Trial of Endobronchial or Endoscopic Ultrasound as a First Test in the Diagnosis and Staging of Lung Cancer
Brief Title: A New Pathway With BronchOscopic or Oesophageal Ultrasound for Lung Cancer Diagnosis and STaging (BOOST)
Acronym: BOOST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: North Middlesex University Hospital (Other); Barnet and Chase Farm Hospitals NHS Trust (Other); The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Principal Investigator, Sam Janes, Reader in Respiratory Medicine, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 07/0156
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Bronchogenic Carcinoma
Keywords: Lung; Cancer; Staging; Endobronchial; Ultrasound; Endoscopic
MeSH Terms: conditions — Carcinoma, Bronchogenic; Neoplasms | interventions — Bronchoscopy; Magnetic Resonance Spectroscopy; Mediastinoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): Control arm: Current practice for diagnosing and staging lung cancer. Most patients with intra-thoracic disease suspected of lung cancer will undergo bronchoscopy (or CT guided biopsy), PET scan and possibly mediastinoscopy.
  Interventions: Procedure: Bronchoscopy, CT-guided biopsy, PET scan, Mediastinoscopy
- A (Experimental): Active arm: A new pathway for the diagnosis and staging of lung cancer with endobronchial (EBUS) or endoscopic ultrasound (EUS) as a first test. If EBUS or EUS is negative the patient will have PET scan +/- mediastinoscopy.
  Interventions: Procedure: Endobronchial or Endoscopic Ultrasound

INTERVENTIONS:
Procedure: Endobronchial or Endoscopic Ultrasound — Patients with anterior mediastinal or subcarinal disease will undergo EBUS. Patients with posterior, subcarinal or AP window disease will undergo EUS. Patients with no mediastinal disease on CT scan will undergo EBUS.
  Other Names: EBUS: Olympus Keymed BF-UC260F-OL8
  Arms: A
Procedure: Bronchoscopy, CT-guided biopsy, PET scan, Mediastinoscopy — Investigations will be determined by the multi-disciplinary team responsible for the patient
  Arms: B

SUMMARY:
In the UK, staging of lung cancer is time consuming (taking on average more than 3 weeks), costly and inaccurate in up to 20% of cases. The investigators wish to determine whether using the newer techniques of endobronchial ultrasound (EBUS) and endoscopic ultrasound (EUS) improves lung cancer staging. The investigators' hypothesis is that EUS (endoscopic ultrasound) or EBUS (endobronchial ultrasound guided transbronchial needle aspirate) as a first test after CT scan in the diagnosis and staging of lung cancer will result in a reduction in the time from first outpatient appointment to treatment decision, a reduction in the total number of scans and investigative operations, fewer outpatient attendances and a reduction in healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients suspected of lung cancer on CT scan
* Written informed consent
* Able to tolerate bronchoscopy and thoracic surgery

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease that makes it undesirable for the patient to participate in the trial
* Any disorder making reliable informed consent impossible
* Patients with extra-thoracic disease, supraclavicular lymphadenopathy or pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Time from first outpatient appointment to decision to treat | 1 - 3 months

SECONDARY OUTCOMES:
The healthcare costs for diagnosing and staging lung cancer | End of study
The number of tests and outpatient visits a patient requires to be diagnosed and staged with lung cancer | 1 - 3 months
The proportion of lung cancer patients that are diagnosed and staged with a single test after CT scan | 1 - 3 months
The time from first outpatient appointment to treatment | 1 - 3 months
The number of futile thoracotomies | 1 - 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Spiro, MD, Principal Investigator — Univeristy College London NHS Trust; Sam Janes, MD PhD, Study Chair — University College, London; Neal Navani, MD, Study Director — University College, London
Locations (4):
- United Kingdom (4):
  - Barnet General Hospital, London
  - North Middlesex University Hospital, London
  - Whittington Hospital NHS Trust, London
  - University College London Hospital NHS Trust, London

REFERENCES:
- [Background] Herder GJ, Verboom P, Smit EF, van Velthoven PC, van den Bergh JH, Colder CD, van Mansom I, van Mourik JC, Postmus PE, Teule GJ, Hoekstra OS. Practice, efficacy and cost of staging suspected non-small cell lung cancer: a retrospective study in two Dutch hospitals. Thorax. 2002 Jan;57(1):11-4. doi: 10.1136/thorax.57.1.11. PMID 11809983
- [Background] Detterbeck FC, Jantz MA, Wallace M, Vansteenkiste J, Silvestri GA; American College of Chest Physicians. Invasive mediastinal staging of lung cancer: ACCP evidence-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):202S-220S. doi: 10.1378/chest.07-1362. PMID 17873169
- [Background] Silvestri GA, Gould MK, Margolis ML, Tanoue LT, McCrory D, Toloza E, Detterbeck F; American College of Chest Physicians. Noninvasive staging of non-small cell lung cancer: ACCP evidenced-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):178S-201S. doi: 10.1378/chest.07-1360. PMID 17873168
- [Background] De Leyn P, Lardinois D, Van Schil PE, Rami-Porta R, Passlick B, Zielinski M, Waller DA, Lerut T, Weder W. ESTS guidelines for preoperative lymph node staging for non-small cell lung cancer. Eur J Cardiothorac Surg. 2007 Jul;32(1):1-8. doi: 10.1016/j.ejcts.2007.01.075. Epub 2007 Apr 19. PMID 17448671
- [Background] Janes SM, Spiro SG. Esophageal endoscopic ultrasound/endobronchial ultrasound-guided fine needle aspiration: a new dawn for the respiratory physician? Am J Respir Crit Care Med. 2007 Feb 15;175(4):297-9. doi: 10.1164/rccm.200609-1390ED. No abstract available. PMID 17277288
- [Background] Navani N, Spiro SG, Janes SM. Mediastinal staging of NSCLC with endoscopic and endobronchial ultrasound. Nat Rev Clin Oncol. 2009 May;6(5):278-86. doi: 10.1038/nrclinonc.2009.39. PMID 19390554
- [Derived] Navani N, Nankivell M, Lawrence DR, Lock S, Makker H, Baldwin DR, Stephens RJ, Parmar MK, Spiro SG, Morris S, Janes SM; Lung-BOOST trial investigators. Lung cancer diagnosis and staging with endobronchial ultrasound-guided transbronchial needle aspiration compared with conventional approaches: an open-label, pragmatic, randomised controlled trial. Lancet Respir Med. 2015 Apr;3(4):282-9. doi: 10.1016/S2213-2600(15)00029-6. Epub 2015 Feb 4. PMID 25660225